CLINICAL TRIAL: NCT01182454
Title: Clinical Test Report for Blood Pressure Meter of CH-658
Status: Completed | Type: Observational
Sponsor: Citizen Systems Japan Co., Ltd. (Industry)
Responsible Party: Makoto Okamoto, Citizen Systems Japan Co., Ltd.
Other Study IDs: Citizen-658
Record Dates: First submitted 2010-08-12; First posted 2010-08-16 (Estimated); Last update posted 2010-08-16 (Estimated); Status verified 2010-08

CONDITIONS: Blood Pressure
Keywords: blood pressure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Blood pressure meter model CH-658 was to be assessed against the standard mercury sphygmomanometer according to the protocol of the ANSI/AAMI SP-10.

ELIGIBILITY:
Inclusion Criteria:

* 96 subjects with a wide range of blood pressure were selected.

Exclusion Criteria:

* Subjects could be taking antihypertensive medication, but excluded in atrial fibrillation or with any sustained arrhythmia.

Ages: 22 Years to 62 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: community sample
Sampling Method: Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2010-01; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Measure accuracy of blood pressure meter CH-658 | 30 minutes
  Measure the accuracy of blood pressure meter model CH-658 against the standard mercury sphygmomanometer according to the protocol of ANSI/AAMI SP-10

CONTACTS AND LOCATIONS:
Locations (2):
- Japan (2):
  - Sone Clinic, Tokyo
  - Sone Clinic, Toyko